CLINICAL TRIAL: NCT05263778
Title: Cholesterol Lowering Via Bempedoic Acid/Ezetimibe, an ACL-Inhibiting Regimen in Acute Coronary Syndrome (CLEAR ACS) Study
Brief Title: Cholesterol Lowering Via Bempedoic Acid/Ezetimibe, an ACL-Inhibiting Regimen in Acute Coronary Syndrome Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1824539
Record Dates: First submitted 2022-02-14; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases; NSTEMI; STEMI
MeSH Terms: conditions — Cardiovascular Diseases; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Bempedoic acid 180 mg/ezetimibe 10 mg
  Interventions: Drug: Bempedoic Acid / Ezetimibe Oral Tablet
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bempedoic Acid / Ezetimibe Oral Tablet — Bempedoic acid 180 mg/ezetimibe 10 mg by mouth once daily for 12 weeks
  Other Names: Nexlizet
  Arms: Intervention
Drug: Placebo — Matching placebo by mouth once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The overall objective of the Cholesterol Lowering via Bempedoic Acid/Ezetimibe, an ACL-Inhibiting Regimen in Acute Coronary Syndrome ACS (CLEAR ACS) study is to determine the efficacy, safety, and tolerability of bempedoic acid/ezetimibe (BA/E) in a contemporary and real-world population, enriched for older adults, women, and underrepresented racial/ethnic groups, of adults with a recent acute coronary syndrome (ACS) event independent of use of statin therapy before the ACS event.

DETAILED DESCRIPTION:
The CLEAR ACS study is a prospective, virtual, electronic health record (EHR)-based, randomized, double-blind, placebo-controlled, parallel-group, pragmatic clinical trial (PCT) embedded within Kaiser Permanente Northern California's fully integrated and learning health care delivery system. The EHR will be screened in real-time for potentially eligible participants across all Kaiser Permanente Northern California hospitals using validated diagnostic and procedural codes, disease registries, laboratory values, pharmacy dispensing information, and sociodemographic data sources. Eligible patients that provide informed consent will be randomized in a 1:1 allocation ratio to an initial 12 weeks of blinded bempedoic acid/ezetimibe (BA/E) vs. matching placebo followed by a 12-week open-label extension phase where all patients will receive open-label, unblinded bempedoic acid/ezetimibe.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age >18 years
* Able to provide informed consent
* A documented recent ACS event (i.e., defined as up to 14 days post-discharge from an index hospitalization for a non-ST-elevation MI [NSTEMI] or ST-elevation MI [STEMI] necessitating urgent and/or emergent percutaneous coronary intervention [PCI] and/or coronary after bypass graft [CABG])
* At least 6 months of continuous health plan membership and prescription drug benefit prior to enrollment
* A registered e-mail address with Kaiser Permanente in order to obtain electronic consent (eConsent) for study participation

Exclusion Criteria:

* Receipt of BA/E on or within 3 months before the day of enrollment
* A history of hypersensitivity to BA/E
* Women who are pregnant or planning to become pregnant and/or breastfeeding mothers
* A diagnosis of gout and/or previously known laboratory-confirmed hyperuricemia (serum uric acid >8.0 mg/dL)
* A history of tendon disorders or tendon rupture
* Current and/or planned treatment with simvastatin/pravastatin, cyclosporine, fibrates, and/or bile acid sequestrants (to avoid drug-drug interactions)
* A known life-limiting diagnosis (e.g., stage D heart failure, severe liver disease, end-stage kidney disease [ESKD] requiring chronic dialysis or an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, metastatic cancer and/or actively receiving systemic chemotherapy)
* Institutionalized and/or receiving palliative care
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of BA/E vs. matching placebo on LDL-C level following a recent ACS event. | 0-12 weeks
  Percent (%) change from baseline to week 12 in LDL-C level

SECONDARY OUTCOMES:
To determine the efficacy of BA/E vs. matching placebo on the lipid profile following a recent ACS event. | 0-12 weeks
  - Percent (%) change from baseline to week 12 in high-density lipoprotein cholesterol (HDL-C)
To determine the efficacy of BA/E vs. matching placebo on the lipid profile following a recent ACS event. | 0-12 weeks
  - Percent (%) change from baseline to week 12 in non-HDL-C
To determine the efficacy of BA/E vs. matching placebo on the lipid profile following a recent ACS event. | 0-12 weeks
  - Percent (%) change from baseline to week 12 in total cholesterol (TC)
To determine the efficacy of BA/E vs. matching placebo on the lipid profile following a recent ACS event. | 0-12 weeks
  - Percent (%) change from baseline to week 12 in triglyceride (TGs) levels

OTHER OUTCOMES:
To assess the safety and tolerability of BA/E vs. matching placebo following a recent ACS event. | 0-12 weeks
  - Proportion (%) of adverse events (AEs) leading to permanent study drug discontinuation and unexpected serious AEs (SAEs) at 12 weeks
To explore the clinical effectiveness of BA/E vs. usual care on all-cause and cause-specific morbidity and mortality following a recent ACS event. | 0-12 weeks
  - Rate (# of events per 100 person-years) of all-cause mortality (ACM)
To explore the clinical effectiveness of BA/E vs. usual care on all-cause and cause-specific morbidity and mortality following a recent ACS event. | 0-12 weeks
  - Rate (# of events per 100 person-years) of MACE (3-point) = death due to any cause, MI, and/or stroke/TIA
To explore the clinical effectiveness of BA/E vs. usual care on all-cause and cause-specific morbidity and mortality following a recent ACS event. | 0-12 weeks
  - Rate (# of events per 100 person-years) of MACE (4-point) = MACE (3-point) + hospitalization for unstable angina
To explore the clinical effectiveness of BA/E vs. usual care on all-cause and cause-specific morbidity and mortality following a recent ACS event. | 0-12 weeks
  - Rate (# of events per 100 person-years) of MACE (5-point) = MACE (4-point) + any coronary revascularization
To explore the clinical effectiveness of BA/E vs. usual care on all-cause and cause-specific morbidity and mortality following a recent ACS event. | 0-12 weeks
  - Rate (# of events per 100 person-years) of all-cause emergency department (ED) visits + all-cause hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Ambrosy, MD, Principal Investigator — Kaiser Permanente Northern California Division of Research; Alan S Go, MD, Principal Investigator — Kaiser Permanente Northern California Division of Research
Locations (1):
- Kaiser Permanente Northern California Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No